CLINICAL TRIAL: NCT00409812
Title: A Double Blinded Randomised Controlled Trial of the Effects of Sodium Citrate on Olfactory Thresholds
Brief Title: A Study of the Effects of Sodium Citrate on Olfactory Thresholds
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospitals, Leicester (Other)
Other Study IDs: 06/MRE05/16
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2007-01-19 (Estimated); Status verified 2007-01

CONDITIONS: Anosmic and Hyposmic Patients

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The study will be undertaken at the ENT department of the Leicester Royal Infirmary and in a research laboratory at the University of Leicester and also in the ENT department at the West Suffolk Hospital. One hundred subjects will be recruited. Subjects will be invited to undergo a series of smell tests using graded concentrations of 4 odours in 120ml bottles (1). This test has been described and validated by our previous work (2). The test will be fully explained to the subject beforehand by the researcher who will test the patient. The subject will be started with the smallest concentration of each odour and will ascend through the bottles until they detect 2 in a row, at which point the weaker concentration of the odour will be taken as their threshold. They will have a threshold levels determined for the odours phenethyl alcohol (roses), mercaptan (gas), acetic acid (vinegar) and eucalyptol (menthol).

Then, the subject will undergo a sodium citrate nasal douche at a specific concentration or will douche with sterile water. There will be three concentrations used (3%, 6% and 9%) and a control solution (sterile water). Patients will be randomly allocated to one of the four groups using a coded bottle system. Both patient and tester will be blinded to the solution used as these will be made in the pharmacy and coded for anonymity - the code will be broken at the end of the trial. Subjects will then be retested with the bottles and threshold levels will be observed for the four odours at 15 minute intervals over 2 hours. The purpose of the repeated tests is to determine the length of the effect (if present) of the citrate on the olfactory ability of the patients.

(N.B. Sodium citrate is a licensed product for use in body cavities (e.g. stomach, bladder) and can be found in the British National Formulary - the concentrations proposed do not exceed those used elsewhere.)

1. Wudarski TJ, Doty RL. Comparison of detection threshold values determined using glass sniff bottles and plastic squeeze bottles.Percept Mot Skills. 2004 Feb;98(1):192-6
2. Gaskin J, Robinson A, Philpott CM, Goodenough P, Murty G. Are patients cross-sensitive to odours in parallel threshold tests? Chemical Senses 2006; in progress

ELIGIBILITY:
Inclusion Criteria:

* Anosmia
* Hyposmia

Exclusion Criteria:

* Under age of 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Julian Gaskin, MBChB MRCSEd, Principal Investigator — University Hospitals, Leicester